CLINICAL TRIAL: NCT03401996
Title: tDCS Over the Supplemental Motor Area for the Treatment of Tourette Syndrome
Brief Title: tDCS in Tourette (TIC-TDCS)
Acronym: TIC-TDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB17-1615
Record Dates: First submitted 2018-01-02; First posted 2018-01-17 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS (Experimental)
  Interventions: Device: 1 mA tDCS over bilateral SMA
- Sham tDCS (Sham Comparator)
  Interventions: Device: 1 mA tDCS over bilateral SMA

INTERVENTIONS:
Device: 1 mA tDCS over bilateral SMA — A 1mA direct current will be delivered through two 5cm x 5cm saline-soaked surface sponge electrodes by a battery-driven, constant-current stimulator (Neuroconn DC stimulator). First, the SMA will be identified based on the guidelines of the international 10-20 electrode system. The tDCS will then be applied using the following procedure:
  1. The head of participants will be measured to find the 'vertex' (top) of the head. This point will be used as a landmark to locate the SMA. This region corresponds to the FCZ (e.g., Legon et al., 2013).
  2. The return electrode will be placed over the mastoids. Once the electrodes are in position, cathodal tDCS will be applied at 1mA for 15 minutes, 2 times a day with a resting period of 20 minutes in between treatment periods, for 5 consecutive days.

SUMMARY:
Double-blind randomized, sham-controlled clinical trial of 1 mA bilateral supplementary motor area in adolescents/adults with Tourette syndrome (TS). The primary objectives are to assess and quantify the safety and efficacy on tic severity of 5 inhibitory sessions of active vs. sham tDCS sessions during active tic suppression, and to explore the differences in brain functional activity before and after 5 sessions of active or sham cathodal tDCS in adolescents and adults with TS. Secondary objectives include the assessment of the severity of comorbidities after 5 inhibitory tDCS sessions.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet Diagnostic and Statistical Manual of Mental Disorders criteria for TS (APA, DSM V).
* 16 years of age or older.
* A "moderately ill" or worse score on the Clinical Global Impression Severity scale (CGI-S).
* A total motor tic or vocal tic severity score greater or equal to 15/25 on the Yale Global Tic Severity Scale (YGTSS) or a combined score greater than 22/50.
* Participants should be either un-medicated or on stable medication treatment for tics for the previous 3 months. If receiving botulinum toxin treatment, their enrolment should be at least 16 weeks after the last treatment session.
* Psychiatric comorbidities should be clinically stable; treatment has not changed in the last 3 months.

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

* Have a metal object/implant in their brain, skull, scalp, or neck.
* Have an implantable device (e.g., cardiac pacemaker).
* Have a diagnosis of epilepsy or cardiac disease.
* Have a history of traumatic brain injury, learning disability or dyslexia.
* Have a severe impediment in vision or hearing.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Tic severity total subscore on the Yale Global Tic Severity Scale (YGTSS) | Immediately after last tDCS session
  The Yale Global Tic Severity Scale is the most extensively deployed scale worldwide for measuring tic severity. It requires an experienced clinician using all available information to rate motor and phonic tic severity during the previous week. Five dimensions (number, frequency, intensity, complexity, and interference) of motor and phonic tics are rated separately on a six point Likert-type scale (zero-five), with each point anchored to descriptive statements and relevant examples. The global score has a zero-one hundred range, composed by severity and overall impairment scores, each of which having a zero-fifty range. Higher values indicate worse outcome.
Tic severity total subscore on the Yale Global Tic Severity Scale (YGTSS) | 1 week after end of intervention
  The Yale Global Tic Severity Scale is the most extensively deployed scale worldwide for measuring tic severity. It requires an experienced clinician using all available information to rate motor and phonic tic severity during the previous week. Five dimensions (number, frequency, intensity, complexity, and interference) of motor and phonic tics are rated separately on a six point Likert-type scale (zero-five), with each point anchored to descriptive statements and relevant examples. The global score has a zero-one hundred range, composed by severity and overall impairment scores, each of which having a zero-fifty range. Higher values indicate worse outcome.

SECONDARY OUTCOMES:
Tic inhibition potential on the Modified Video-Based Tic Rating Scale (MVBTRS) | Immediately after and 1 week after last tDCS session
  Tic suppression will be measured using the Modified Rush Video-Based Tic Rating Scale through a 5 min video recording (2.5 min head and shoulders and 2.5 min whole body view). The scoring method consists of combining scores rating tic distribution (number of body areas involved, from 0 to 4), tic frequency (number of motor and phonic tics expressed from 0 to 4), and tic severity (for motor tics and for phonic tics, from 0 to 4). The total score range is 0 to 20, with higher values indicating worse outcome. Tic suppression will be expressed as suppression potency (IP), defined as follows: IP = RF-RI/RF, where RF is the Rush score during 'free' ticcing and RI the Rush score during tic suppression. Thus, the higher the IP value, the more efficient the suppression potency.
Adverse effects | Immediately after and 1 week after last tDCS session
  Semistructured questionnaire on adverse effects
Tourette Syndrome Clinical Global Impression (TS-CGI) | Immediately after and 1 week after last tDCS session
  The TS-CGI is a clinician-rated seven point ordinal scale that ranks current symptom severity from "normal" to "extremely severe", rating the overall adverse impact of tics, but does not assess separately the individual dimensions of tics. It shares the same composition with Clinical Global Impression of Severity scales, which are commonly used measures of symptom severity in studies of patients with psychiatric disorders.
Individualized-Premonitory Urge for Tics Scale (iPUTS) | Immediately after and 1 week after last tDCS session
  The I-PUTS is a clinician-administered measure that assessed the presence, frequency, intensity, and body region location of urges for individual tics endorsed over the past week using a symptom checklist that paralleled the YGTSS. The clinician inquires about the frequency of endorsed urges on a 4-point scale (1 = "Urge occurs 0-25% of the time you do the tic" to 4 = "Urge occurs 75%-100% of the time you do the tic"). The clinician also inquires about the urge intensity on a 4-point scale (1 = "minimal intensity/urge can be ignored for a considerable amount of time" to 4 = "strong intensity/urge needs relief almost immediately"). When tics and/or urges are not endorsed, items receive a rating of 0. Finally, the clinician inquires about the body region associated with each urge. Items are summed to create a total number of distinct urges (I-PUTS Urge Number), total urge frequency (I-PUTS Frequency), and total urge intensity (I-PUTS Intensity).
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Immediately after and 1 week after last tDCS session
  The Y-BOCS is a 10-item, clinician-administered scale, that has become the most widely used rating scale for obsessive-compulsive disorder. The Y-BOCS provides five rating dimensions for obsessions and compulsions: time spent or occupied; interference with functioning or relationships; degree of distress; resistance; and control (i.e., success in resistance). The 10 Y-BOCS items are each scored on a four-point scale from 0 = "no symptoms" to 4 = "extreme symptoms." The sum of the first five items is a severity index for obsessions, and the sum of the last five an index for compulsions. A translation of total score into an approximate index of overall severity ranges between 0 and 40, with higher scores indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Davide Martino, MD, PhD, Principal Investigator — Department of Clinical Neurosciences, University of Calgary
Locations (1):
- Department of Clinical Neurosciences, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No